CLINICAL TRIAL: NCT03838679
Title: Multimodal Imaging of Subretinal Fibrosis in Neovascular AMD
Brief Title: Imaging of the Angiofibrotic Switch in Neovascular AMD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Philipp Roberts, Principal investigator, Medical University of Vienna
Other Study IDs: 2019-02-0051
Record Dates: First submitted 2019-02-10; First posted 2019-02-12 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Age-related Macular Degeneration; Choroidal Neovascularization
MeSH Terms: conditions — Macular Degeneration; Choroidal Neovascularization | interventions — Tomography, Optical Coherence; Fluorescein Angiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: 80 participants with neovascular AMD and a minimum history of 12 months of anti- VEGF therapy will be included in cohort 1 and examined only once (1 study visit).
  Interventions: Diagnostic Test: Best-corrected Visual acuity testing (BCVA); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Color fundus photography (CFP); Diagnostic Test: Optical coherence tomography angiography (OCTA); Diagnostic Test: Polarization-sensitive optical coherence tomography (PS-OCT); Diagnostic Test: Microperimetry (MP); Diagnostic Test: Adaptive-optics optical coherence tomography (AO-OCT); Diagnostic Test: Fluorescein angiography (FA)
- Cohort 2: 40 participants with treatment-naive neovascular AMD receiving standardized anti- VEGF therapy will be included in cohort 2 and followed for 12 months (6 study visits).
  Interventions: Diagnostic Test: Best-corrected Visual acuity testing (BCVA); Diagnostic Test: Optical coherence tomography (OCT); Diagnostic Test: Color fundus photography (CFP); Diagnostic Test: Optical coherence tomography angiography (OCTA); Diagnostic Test: Polarization-sensitive optical coherence tomography (PS-OCT); Diagnostic Test: Microperimetry (MP); Diagnostic Test: Adaptive-optics optical coherence tomography (AO-OCT); Diagnostic Test: Fluorescein angiography (FA)

INTERVENTIONS:
Diagnostic Test: Best-corrected Visual acuity testing (BCVA) — Best-corrected visual acuity (BCVA) will be measured using Early Treatment of Diabetic Retinopathy Study (ETDRS) charts at 4 meters and 1 meter, respectively.
Diagnostic Test: Optical coherence tomography (OCT) — Optical Coherence Tomography (OCT) is a non-invasive diagnostic technique that renders an in vivo cross sectional view of the retina.
Diagnostic Test: Color fundus photography (CFP) — Color fundus photography is a non-invasive, fast and reliable imaging method providing a true-to-life depiction of the ocular fundus.
Diagnostic Test: Optical coherence tomography angiography (OCTA) — OCTA, an extension of conventional OCT, offers noninvasive imaging of the retinal and choroidal vasculature.
Diagnostic Test: Polarization-sensitive optical coherence tomography (PS-OCT) — PS-OCT, a functional exten- sion of conventional OCT technology, enables differentiation of retinal layers based on their distinct interference with the polarization state of the probing light beam, as opposed to mere light intensity.
Diagnostic Test: Microperimetry (MP) — Microperimetry allows testing of retinal sensitivity at specific locations in the area of the fovea, parafovea or even more peipheral areas of the macula.
Diagnostic Test: Adaptive-optics optical coherence tomography (AO-OCT) — AO-OCT, an extension of conventional OCT, offers non-invasive imaging of the retina with improved lateral resolution of up to 2-3 μm.
Diagnostic Test: Fluorescein angiography (FA) — FA imaging is a standard imaging technique used for the diagnosis of vascular pathologies of the retina such as choroidal neovascularization.

SUMMARY:
The content of this research project is to identify the angiofibrotic switch, the transition from angiogenesis to fibrosis, in neovascular age-related macular degeneration (nAMD) longitudinally. Despite optimal treatment about 50% of eyes with nAMD develop fibrosis within 2 years, causing irreversible damage to the retina and functional loss. Objective measurement of fibrosis, however, is challenging, since clinical staging is subjective and current imaging modalities such as color fundus photography (CFP), fluorescein angiography (FA) and optical coherence tomography (OCT) often do not allow clear delineation. Novel imaging modalities such as polarization-sensitive OCT (PS-OCT), OCT angiography (OCTA) and adaptive-optics OCT (AO-OCT) offer identification of fibrous components and microvasculature of fibrotic lesions non-invasively with highest precision and shall thus be used in this study.

Hypotheses: The investigators hypothesize to detect and quantify subclinical (i.e. not detectable on dilated fundus examination) areas of fibrosis using PS-OCT and determine the rate and exact location within the neovascular lesion. Furthermore, the investigators expect neuroretinal and microvascular changes, which will be assessed by AO-OCT and OCTA.

Methods: Eighty eyes of 80 patients with chronic nAMD will be included and examined cross- sectionally to evaluate the accuracy of PS-OCT to detect and quantify fibrosis in comparison to gold standard imaging modalities. In addition, OCTA and AO-OCT will be performed to analyze the relationship between fibrous, neovascular and neuroretinal structures. Furthermore, forty eyes of 40 participants with treatment-naïve nAMD will be included and followed over 12 months with predefined follow-up intervals. Novel non-invasive imaging will be applied to objectively determine the exact time and extent of the angiofibrotic switch in nAMD during state-of-the- art therapy. This approach has not been done before and is clinically relevant for multiple reasons: Firstly, only little is known about the development of fibrosis in AMD during therapy. Secondly, the clinical diagnosis of subretinal fibrosis is subjective and does not allow reliable quantification. Thirdly, current gold standard imaging modalities (i.e. CFP and FA) for detection of fibrosis involve invasive and time-consuming procedures and do not allow three-dimensional analysis. Finally, our study may identify objective endpoints for future interventional trials.

DETAILED DESCRIPTION:
Research questions/hypotheses: Age-related macular degeneration (AMD) is the main cause of legal blindness among elderly patients in industrialized countries. The main reason for severe and irreversible visual impairment among these patients is subretinal fibrosis (SF). Large-scale interventional trials (e.g. CATT) have shown that half of all eyes affected by choroidal neovascularization (CNV) develop clinically visible fibrotic scarring over two years despite optimal treatment, causing irreversible retinal damage and functional loss. Thus, prevention of fibrosis in AMD is currently the focus of researchers worldwide. Clearly defined end points for interventional trials, however, are lacking because detection and quantification of SF is challenging. Clinical staging of SF is subjective and current gold standard imaging modalities such as color fundus photography (CFP), fluorescein angiography (FA) and optical coherence tomography (OCT), even in concert, do not allow a distinct and early delineation of SF. Novel imaging modalities such as polarization-sensitive OCT (PS-OCT), OCT angiography (OCTA) and adaptive optics (AO)-OCT are promising means to objectively detect SF and provide detailed insights into the biology of the microvascular and neurosensory compartments. Our group recently demonstrated that PS-OCT offers automated identification and quantification of SF in AMD based on tissue-specific contrast. Aim of the proposed research project is to detect and characterize the angiofibrotic switch, i.e. the transition from active and reversible neovascularization to irreversible fibrosis, in neovascular AMD under anti-VEGF treatment. We hypothesize to detect the initiating events of fibrotic conversion including even subclinical stages of fibrosis by non-invasive PS-OCT and identify the association with fibrovascular and retinal changes by OCTA and AO-OCT, respectively.

Scientific/scholarly innovation/originality of the project: The combination of PS-OCT, OCTA and AO-OCTA to non-invasively detect pathognomonic features of fibrovascular conversion is a novel and unprecedented approach towards objective visualization and quantification of disease pathomechanisms. Outcomes of this study may provide clearly defined morphological endpoints for future interventional trials.

Methods: Eighty eyes of 80 patients with chronic nAMD will be included and examined cross-sectionally to evaluate the accuracy of PS-OCT to detect and quantify fibrosis in comparison to gold standard imaging. In addition, OCTA and AO-OCT will be performed to analyze the relationship between fibrous, vascular and retinal structures. Furthermore, forty eyes of 40 participants with treatment-naïve nAMD will be included in a prospective study and followed for one year under treatment. PS-OCT, AO-OCT and OCTA imaging will be performed according to a standardized protocol at predefined visits. Gold standard imaging will be performed for validation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neovascular AMD with anti-VEGF treatment of a minimum duration of 12 months (cohort 1)
* Treatment-naïve active neovascular AMD (cohort 2)
* 50 years of age or older
* Visual acuity 20/25-20/320
* At least one druse (>63μm) in either eye or late AMD in the fellow eye
* Fibrosis <50% of total lesion area at baseline (cohort 2)

Exclusion Criteria:

* Previous treatment for CNV in the study eye (cohort 2)
* Presence of other progressive retinal disease likely to affect visual acuity
* Contraindications for treatment with anti-VEGF
* Pregnancy
* Dyslexia

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: There will be two study cohorts in this trial:
  1. 80 participants with neovascular AMD and a minimum history of 12 months of anti- VEGF therapy will be included in cohort 1 and examined only once (1 study visit).
  2. 40 participants with treatment-naive neovascular AMD receiving standardized anti- VEGF therapy will be included in cohort 2 and followed for 12 months (6 study visits).
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-04-28 (Estimated); Study Completion 2022-04-28 (Estimated)

PRIMARY OUTCOMES:
Detection of subretinal fibrosis by PS-OCT | 15 months
  The primary objective is to determine how well the fibrosis present/not present classification of the novel PS-OCT imaging works compared to gold standard imaging techniques. To assess the primary objective, a 95% confidence interval for the proportion of correct fibrosis yes/no classifications by the novel PS-OCT imaging compared to the gold standard will be computed. To assess this objective, data from cohort 1 will be used.

SECONDARY OUTCOMES:
Extension of fibrosis area quantified on PS-OCT and correlated to standard imaging modalities | 33 months
  The secondary objective is to determine how well the fibrosis area detection of the novel PS-OCT imaging works compared to gold standard imaging techniques. To assess the secondary objective, a Bland-Altman plot will be drawn. Furthermore, a 95% confidence interval for the mean difference in detected area and the mean absolute difference in detected area will be computed. To assess this objective, two analysis sets will be used: Firstly, data from cohort 1 and baseline data of cohort 2, and secondly data from the 1 year follow-up examination of patients in cohort 2.

OTHER OUTCOMES:
Correlation of fibrosis and co-localized vascular changes (comparison between OCTA and PS-OCT) | 36 months
  In cohort 1 (eyes with a minimum history of 12 months of anti- VEGF), we will compare imaging data assessed by PS-OCT with image data from OCTA for morphological analyses. In cohort 2 the same analyses will be performed. Cohort 2 will provide detailed follow-up information about morphological changes over time. Outcome measures in eyes with and without fibrosis (vessel configuration in OCTA) will be compared using chi-square tests (categorical variables), t-tests (metric variables that can be assumed to be normally distributed) and Wilcoxon tests (metric variables that cannot be assumed to be normally distributed). ANOVA and paired t-tests will be used to investigate the longitudinal changes in cohort 2. P values < 0.05 will be considered statistically significant. Due to the exploratory nature of these analyses, no correction for multiplicity will be used.
Correlation of fibrosis localization and co-localized retinal function (comparison between MP, PS-OCT, OCTA, OCT and AO-OCT) | 36 months
  For a morphological-functional analysis areas of functional loss in microperimetry will be analyzed in detail using multimodal imaging (including PS-OCT, OCTA, OCT and AO-OCT) and relevant morphological changes associated with reduced retinal sensitivity will be assessed and described. In cohort 1 and cohort 2 the same analyses will be performed. Additionally, cohort 2 will provide detailed follow-up information about morphological and functional changes over time.
Correlation of morphology (fibrosis) and visual outcome (comparison between BCVA and PS-OCT, OCTA, AO-OCT, OCT) | 36 months
  Descriptive analysis will be performed for patient demographics of both cohort 1 and cohort 2, as well as for morphological parameters and visual acuity (for metric variables mean, standard deviation, min, max, median and for categorical variables absolute and relative frequencies will be computed). Outcomes of BCVA testing in eyes with and without subretinal fibrosis will be analyzed cross-sectionally (cohort 1) and longitudinally (cohort 2).
Condition of the retinal pigment epithelium (RPE) assessed by PS-OCT in areas of fibrosis. | 36 months
  Condition of the RPE assessed by PS-OCT will be graded as continuous, RPE porosity, focal RPE atrophy, RPE thickening or pigment migration in areas with and without fibrosis and described. RPE condition in eyes with and without subretinal fibrosis will be analyzed cross-sectionally (cohort 1) and longitudinally (cohort 2).
Correlation of fibrosis localization and co-localized photoreceptor status (comparison between AO-OCT and PS-OCT) | 36 months
  Condition of the photoreceptor layer assessed by AO-OCT in areas with and without fibrosis (particularly areas at the border zone of subretinal fibrosis) will be assessed and described. RPE condition in eyes with and without subretinal fibrosis will be analyzed cross-sectionally (cohort 1) and longitudinally (cohort 2).

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Roberts, MD PhD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided